CLINICAL TRIAL: NCT06848270
Title: Effectiveness of Early Intervention in Palliative Care for Acute Myeloid Leukemia Patients Comparing to Standard of Care: a Randomized Pragmatic Clinical Trial, 1:1 Ratio, Parallel Group and Superiority Study
Brief Title: Effectiveness of Early Intervention in Palliative Care for Acute Myeloid Leukemia Patients Comparing to Standard of Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Acute myeloid leukemia
Record Dates: First submitted 2025-02-03; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Palliative Care; Acute Myeloid Leukaemia
Keywords: Acute myeloid leukaemia; Palliative care
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Randomized pragmatic clinical trial, 1:1 ratio, parallel group and superiority study that compares the effectiveness of early intervention of palliative care in acute myeloid leukemia patients comparing to standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early follow up by the palliative care team (Active Comparator): Early follow up by the palliative care team, that is, from diagnosis
  Interventions: Other: Early palliative care integration
- Standard of care: conventional treatment (No Intervention): Conventional treatment by the Hematology team where this referral is made only in specific cases in which hematologists understand that this need exists.

INTERVENTIONS:
Other: Early palliative care integration — Early follow up by the palliative care team, from diagnosis
  Arms: Early follow up by the palliative care team

SUMMARY:
Hemato-oncology patients undergoing intensive chemotherapy treatments experience different types of symptoms during and after treatments, which are often refractory to the established therapy. Physical symptoms such as pain, dyspnea, mucositis, insomnia, loss of appetite, constipation and diarrhea, among others, have a huge impact on quality of life, temporarily until symptomatic control, but also permanently with the development of anxiety, depression, long-term fatigue and post-traumatic stress. As recommended by ASCO (American Society of Clinical Oncology), the palliative approach to oncological diseases must be as early as possible and be part of the "standard of care". However, the lack of concrete data on this topic in the last decade served as a barrier to the early integration of this same care for hemato-oncology patients in its various areas. Palliative care presupposes global, interdisciplinary action, carried out by specific teams that must act in situations of incurable or serious illness, in an advanced and progressive phase. The potential benefits can be countless and of significant importance, from the impact on quality of life, symptomatic control, reduction of anxiety and depression and even the promotion of informed and conscious choices at the end of life as well as the reduction of aggressive strategies. used at this stage of the disease.

DETAILED DESCRIPTION:
Hematological diseases are biologically complex and constitute a group of oncological pathologies in which the acute disease has an unpredictable course and can reach different outcomes quickly. Patients often experience rapid and not always predictable progression during their treatment trajectory and at the end of life. Unlike most advanced solid tumors, the possibility of cure remains an objective even in situations of relapse or refractory disease. Hemato-oncology patients undergoing intensive chemotherapy treatments experience different types of symptoms during and after treatments, which are often refractory to the established therapy. Physical symptoms such as pain, dyspnea, mucositis, insomnia, loss of appetite, constipation and diarrhea, among others, have a huge impact on quality of life, temporarily until symptomatic control, but also permanently with the development of anxiety, depression, long-term fatigue and post-traumatic stress. As recommended by ASCO (American Society of Clinical Oncology), the palliative approach to oncological diseases must be as early as possible and be part of the "standard of care". However, the lack of concrete data on this topic in the last decade served as a barrier to the early integration of this same care for hemato-oncology patients in its various areas. There are still many specific needs that have not been identified, especially in the initial approach to acute illness. Palliative care presupposes global, interdisciplinary action, carried out by specific teams that must act in situations of incurable or serious illness, in an advanced and progressive phase. The palliative approach can begin with palliative actions carried out by professionals without specific training so that, in inpatient or outpatient settings, the negative repercussions of the disease can be reduced on the various aspects of the patient: physical, psychological, social and spiritual. To this end, palliative interventions must be developed and defined based on the greatest needs of this population and the timing of the disease, not just at the end of life. The potential benefits can be countless and of significant importance, from the impact on quality of life, symptomatic control, reduction of anxiety and depression and even the promotion of informed and conscious choices at the end of life as well as the reduction of aggressive strategies. used at this stage of the disease.

The still scarce knowledge among hematologists about the benefits of palliative care in this population has represented an important barrier. In intensive chemotherapy, area of palliative care that have been little intervened, there seems to be an enormous potential for benefit with these interventions given the complexity of physical and psychological symptoms involved, with "cure" being the main objective. Our aim is to evaluate the effect of early follow-up by the palliative care team compared to conventional treatment by the Hematology team, where this referral is made only in specific cases.

ELIGIBILITY:
Inclusion Criteria:

* Capable of making decisions
* Diagnosed with acute myeloid leukemia
* Aged 70 years or less
* Treated or referred for treatment at the Hematology department of Centro Hospitalar e Universitário de São João.

Exclusion Criteria:

* All patients referred for "best supportive care", that is, for supportive care including treatment with cytoreductive intent.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue | At diagnosis/start of treatment; After induction cycle (approximately after 1 month); After consolidation cycles (approximately after 2 and 3 months)
  Assessment of participant fatigue using the Fatigue Scale FACIT. The lower the score, the higher the fatigue.
Quality of life - Functional Scale, Global Health Status, Symptom Scale | At diagnosis/start of treatment; After induction cycle (approximately after 1 month); After consolidation cycles (approximately after 2 and 3 months)
  Assessment of quality of life using the questionnaire EORTC QLQ-C30. Contains 30 questions assessing three dimensions: 1) Functional Scales: The higher the score, the greater the functional level. 2) Global Health Status: The higher the score, the better the quality of life. 3) Symptom Scales: The higher the score, the greater the severity or frequency of symptoms.
Anxiety and depression | At diagnosis/start of treatment; After induction cycle (approximately after 1 month); After consolidation cycles (approximately after 2 and 3 months)
  Assessment of anxiety and depression using HADS (Hospital Anxiety and Depression Scale), composed of two subscales for anxiety and depression, each with scores categorized as normal (0-7), mild (8-10), moderate (11-14), and severe (15-21). A score ≥ 11 indicates the presence of anxiety and/or depression.
Symptoms and multidimensional well-being | At diagnosis/start of treatment; After induction cycle (approximately after 1 month); After consolidation cycles (approximately after 2 and 3 months)
  Assessment of symptoms and multidimensional well-being using the scale IPOS (Palliative care Outcome Scale). Composed by: Q1: Open-ended question, no scoring, used to guide care; Q2-Q5: Scales of 0-4, where higher scores indicate greater symptom severity; Q6-Q8: Positive items, scored 0-4, where lower scores are better; Q10: Open-ended question, no scoring. Sum of the scores from the rated questions (0-68).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar e Universitário de São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No